CLINICAL TRIAL: NCT05761184
Title: Characterization of Serum Proteome in Subjects Suffering From Prader Willi Syndrome With Different Degrees of Liver Steatosis
Brief Title: Characterization of Serum Proteome in Subjects With Prader Willi Syndrome (PROTEOMARKER)
Acronym: PROTEOMARKER
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C216
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-03

CONDITIONS: Prader-Willi Syndrome
Keywords: Obesity; Genetic obesity; Biomarkers; Proteoma
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steatosis grade 2-3: Subjects with Prader-Willi syndrome and with steatosis grade 2-3
  Interventions: Diagnostic Test: Serum collection for proteomic analysis
- Steatosis grade 0-1: Subjects with Prader-Willi syndrome and with steatosis grade 0-1
  Interventions: Diagnostic Test: Serum collection for proteomic analysis

INTERVENTIONS:
Diagnostic Test: Serum collection for proteomic analysis — Serum collection for proteomic analysis

SUMMARY:
The lack of serum markers that can be used to identify the levels of steatosis in obese subjects, or that can indicate a rapid progression of the metabolic disease, in which it is very often difficult to perform analyzes with imaging techniques, limits the current evolution from a generalized medicine to a personalized medicine. With the project proposal the aim is to identify serum markers for the characterization of steatosis in subjects affected by genetic obesity, which will most likely also be used in metabolic obesity.

DETAILED DESCRIPTION:
Methods Study design The study includes two phases, a first exploratory phase known as "discovery" in which 30 subjects with Prader-Willi Syndrome (PWS) will be analyzed with SOMAscan technology to perform a serum proteomic profile. Hepatic steatosis will be determined by the use of abdominal ultrasound in PWS subjects by establishing the control group (steatosis grade 0/1) and the steatotic one (steatosis grade 2/3). Subsequently, at least two candidate biomarkers will be selected and validated by ELISA in the 30 samples used in the discovery phase (samples already present in our serum bank) and a further 22 samples from PWS patients specifically enrolled for this study.

Patients:

30 subjects already recruited in our previous MIRNOMAPWS project (RC-2018) with genetic diagnosis of PWS, of both sexes and aged between 18 and 45 years in baseline conditions, will be taken into consideration.

For each patient, the following variables will be collected from the medical records:

* anthropometric parameters (height, weight, BMI, waist circumference);
* body composition (lean mass, fat mass), using the impedance measurement technique (BIA);
* levels of steatosis measured with ultrasound according to standard criteria
* basic metabolism, using indirect calorimetry;
* biochemical parameters determining the metabolic syndrome (HDL cholesterol, triglycerides, blood sugar);
* blood pressure;
* concomitant hormonal therapies (growth hormone therapy, sex steroids, and/or l-thyroxine).

Serum collection for proteomic analysis: the proteomic analysis will be performed on the 30 samples already available (used for the "discovery" phase) and on 22 new patients. Similarly to what was done for the MIRNOMAPWS project (RC-2018), fasting blood samples from new patients will be collected by standard venipuncture in BD Vacutainer® serum separation tubes (BD - Plymouth PL6 7BP, UK) and centrifuged at 1900g at 4°C for 10 min and at 16,000 g at 4°C for a further 10 minutes. The supernatants were frozen at -80°C for long-term storage.

Proteomic analysis: before the proteomic analysis the presence of hemoglobin will be evaluated by spectrophotometer Beckman Coulter® DU®730 (Beckman Coulter, Brea, CA, USA) using the direct spectrophotometric method of Harboe with Allen correction: Hb (g / L) = (167, 2 × A415 - 83.6 × A380 - 83.6 × A450) x 1/1000 × 1 / dilution in dH2O. The cut-off considered for serum will be 0.020 g/L.

For the proteomic characterization of serum, a new high-throughput omics technology based on the SomaLogic SOMAscan platform will be used. The system is based on the detection of SOMAmers (Slow Off-rate Modified Aptamers), which are aptameric forms of DNA with high affinity and specificity for the protein target. Furthermore, these aptamers are resistant to nucleotidase activity and demonstrate higher affinity than normal antibodies. The panel used in this study will allow us to evaluate 1500 protein targets that are involved in the development of metabolic diseases, are part of the general inflammatory response, and are of interest in the study of cardiovascular diseases and oncology.

In general, the sensitivity and performance of the test are comparable to that of a normal ELISA kit, with limits for quantification around 100 fM and detection of 40 fM, and the need for only 65 µL of the sample.

Validation of candidates by ELISA: in this phase, at least two of the markers will be validated, identified in the discovery phase, which have demonstrated a significant association with the increase in steatosis in multi-parametric correlation analyses. The validation will be done by quantifying the candidates in the serum samples using specific sandwich-type commercial ELISA kits. As mentioned in the previous section, a total of 52 samples will be measured, 30 of which enrolled for the discovery phase (sera already stored) and another 22 new samples from subjects enrolled for the validation phase.

ELIGIBILITY:
Inclusion Criteria: i. patients with a genetic diagnosis of Prader-Willi syndrome; ii. age range 18-45 years

Exclusion Criteria: i. age < 18 and > 45 years

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients with Prader-Willi syndrome
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Characterization of serum proteome | Baseline
  Evaluation of 1500 protein targets that are involved in the development of metabolic diseases

SECONDARY OUTCOMES:
Relationships with basal resting energy expenditure | Baseline
  Relationships of protein targets with basal resting energy expenditure
Relationships with body composition parameters (evaluated throughout bioimpedentiometry) | Baseline
  Relationships with fat mass and fat free mass

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy